CLINICAL TRIAL: NCT02697916
Title: Aspirin Dosing: A Patient-Centric Trial Assessing Benefits and Long-term Effectiveness
Brief Title: Aspirin Dosing: A Patient-Centric Trial Assessing Benefits and Long-term
Acronym: ADAPTABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Medidata Solutions (Industry); Chicago Area Patient-Centered Outcomes Research Network (CAPriCORN) (Other); Greater Plains Collaborative Clinical Data Research Network (Other); Mid-South Clinical Data Research Network (Other); Research Action for Health Network (REACHnet) (Other); The Patient-Oriented Scalable National Network for Effectiveness Research (Other); PaTH Clinical Data Research Network (Other); New York City Clinical Data Research Network (Other); The Health eHeart Alliance (Other); OneFlorida Clinical Data Research Network (Network); HealthCore-Anthem Research Network (Other); Humana Inc. (Industry); The Patient-Centered Network of Learning Health Systems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00068525
Record Dates: First submitted 2016-02-18; First posted 2016-03-03 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: aspirin; ACSD; PCORI
MeSH Terms: conditions — Atherosclerosis | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- ASA 81mg (Active Comparator): aspirin 81mg
  Interventions: Drug: aspirin
- ASA 325mg (Active Comparator): aspirin 325mg
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: aspirin — 81mg of aspirin daily vs. 325mg of aspirin daily
  Other Names: ASA

SUMMARY:
ADAPTABLE is a pragmatic clinical trial in which 15,000 patients who are at high risk for ischemic events will be randomly assigned in a 1:1 ratio to receive an aspirin dose of 81 mg/day vs. 325 mg/day. Study participants will be enrolled over 38 months. Maximum follow-up will be 50 months. The purpose of the study is to identify the optimal dose of aspirin for secondary prevention in patients with Atherosclerotic cardiovascular disease (ASCVD). The primary endpoint is a composite of all-cause death, hospitalization for MI, or hospitalization for stroke. The primary safety endpoint is hospitalization for major bleeding with an associated blood product transfusion.

DETAILED DESCRIPTION:
In this pragmatic, patient-centered clinical trial, the investigators will compare the effectiveness of two doses of aspirin (81 mg and 325 mg) currently in widespread use in the United States in the secondary-prevention population of patients with established ASCVD. The trial will use a novel format that uses existing electronic health records (EHRs), as well as a web-based patient portal to collect patient-reported outcomes (PROs), and available patient encounter data to supplement/support the EHR. Patients who are identified as candidates for the trial will be directed to the electronic patient portal for the eConsent as well as an abbreviated eligibility confirmation and randomization. One of the important aims of ADAPTABLE is to engage patients, their healthcare providers, and trial investigators in using the infrastructure PCORnet has developed and continues to refine. A total of 15,000 high-risk patients with ASCVD will be randomly assigned (in an open-label fashion) in a 1:1 ratio to instructions to use a daily aspirin dose of either 81 mg or 325 mg daily. The investigators expect the entire sample of patients will be enrolled over 38 months, with a maximum follow-up of 50 months.

ELIGIBILITY:
Inclusion Criteria:

* Known atherosclerotic cardiovascular disease (ASCVD), defined by a history of prior myocardial infarction, prior coronary angiography showing ≥75% stenosis of at least one epicardial coronary vessel, or prior coronary revascularization procedures (either PCI or CABG), or history of chronic heart disease, CAD, ASCVD
* Age ≥ 18 years
* No known safety concerns or side effects considered to be related to aspirin, including
* No history of significant allergy to aspirin such as anaphylaxis, urticaria, or significant gastrointestinal intolerances
* No history of significant GI bleed within the past 12 months
* Significant bleeding disorders that preclude the use of aspirin
* Access to the Internet. In the event that the CDRNs are notified that a cohort of patients without internet access can be included, then patient agreement will be obtained during the consent process to provide follow-up information by telephone contact with the DCRI Call Center.
* Not currently treated with an oral anticoagulant - either warfarin or a novel anticoagulant (dabigatran, rivaroxaban, apixaban, edoxaban) - and not planned to be treated in the future with an oral anticoagulant for existing indications such as atrial fibrillation, deep venous thrombosis, or pulmonary embolism.
* Not currently treated with ticagrelor and not planned to be treated in the future with ticagrelor.
* Female patients who are not pregnant or nursing an infant
* Estimated risk of a major cardiovascular event (MACE) > 8% over next 3 years as defined by the presence of at least one or more of the following enrichment factors:
* Age > 65 years
* Serum creatinine > 1.5 mg/dL
* Diabetes mellitus (Type 1 or Type 2)
* 3-vessel coronary artery disease
* Cerebrovascular disease and/or peripheral arterial disease
* Left ventricular ejection fraction (LVEF) < 50%
* Current cigarette smoker
* Chronic systolic or diastolic heart failure
* SBP > 140 (within past 12 mos)
* LDL > 130 (within past 12 mos)

Exclusion Criteria:

* There will be no exclusions for any upper age limit, comorbid conditions, or concomitant medications other than oral anticoagulants and ticagrelor that are used at the time of randomization, or are planned to be used during the study follow-up.
* Patients and sites interested in participating must be part of the listed health systems collaborators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15076 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William S. Jones, MD, Principal Investigator — Duke Clinical Research Institute; Adrian F. Hernandez, MD MHS FAHA, Principal Investigator — Duke Clinical Research Institute
Locations (40):
- United States (40):
  - UCLA Medical Center, Los Angeles, California
  - HealthCore, Wilmington, Delaware
  - University of Florida Cardiology - Springhill, Gainesville, Florida
  - Florida Hospital, Orlando, Florida
  - Orlando Health, Orlando, Florida
  - Bond Community Health Center, Tallahassee, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Health System, New Orleans, Louisiana
  - Tulane University Heart & Vascular Institute, New Orleans, Louisiana
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Essentia Health St. Mary's Medical Center, Duluth, Minnesota
  - Allina Health, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New York University School of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medicine of Cornell University, New York, New York
  - Montefiore Medical Center, New York, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State Univerity, Columbus, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Baylor Scott and White Heart and Vascular Hospital, Dallas, Texas
  - University of Texas-Southwestern, Dallas, Texas
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - Marshfield Clinic, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Narcisse DI, Whittle J, Rhodes GM, Stebbins AL, Wruck LM, Mulder H, Kripalani S, Munoz D, Effron MB, Gupta K, Handberg EM, Girotra S, Hess R, Benziger CP, Farrehi P, VanWormer JJ, Knowlton KU, Polonsky TS, Bradley SM, Robertson HR, Hammill BG, Rothman RL, Harrington RA, Jones WS, Hernandez AF. Association of study visit interval length with follow-up completeness and adherence to assigned study drug dose: A randomized comparison of participants in the ADAPTABLE trial. Contemp Clin Trials. 2025 Sep;156:108030. doi: 10.1016/j.cct.2025.108030. Epub 2025 Jul 25. PMID 40716702
- [Derived] Marquis-Gravel G, Mulder H, Wruck LM, Benziger CP, Effron MB, Farrehi PM, Girotra S, Gupta K, Kripalani S, Munoz D, Polonsky TS, Whittle J, Harrington R, Rothman R, Hernandez AF, Jones WS. Impact of aspirin dose according to race in secondary prevention of atherosclerotic cardiovascular disease: a secondary analysis of the ADAPTABLE randomised controlled trial. BMJ Open. 2024 Aug 7;14(8):e078197. doi: 10.1136/bmjopen-2023-078197. PMID 39117415
- [Derived] Benziger CP, Stebbins A, Wruck LM, Effron MB, Marquis-Gravel G, Farrehi PM, Girotra S, Gupta K, Kripalani S, Munoz D, Polonsky TS, Sharlow A, Whittle J, Harrington RA, Rothman RL, Hernandez AF, Jones WS. Aspirin Dosing for Secondary Prevention of Atherosclerotic Cardiovascular Disease in Male and Female Patients: A Secondary Analysis of the ADAPTABLE Randomized Clinical Trial. JAMA Cardiol. 2024 Sep 1;9(9):808-816. doi: 10.1001/jamacardio.2024.1712. PMID 38985488
- [Derived] Girotra S, Stebbins A, Wruck L, Marquis-Gravel G, Gupta K, Farrehi P, Benziger CP, Effron MB, Whittle J, Munoz D, Kripalani S, Anderson RD, Jain SK, Polonsky TS, Ahmad FS, Roe MT, Rothman RL, Harrington RA, Hernandez AF, Jones WS. Aspirin Dosing for Secondary Prevention of Atherosclerotic Cardiovascular Disease in Patients Treated With P2Y12 Inhibitors. J Am Heart Assoc. 2023 Oct 17;12(20):e030385. doi: 10.1161/JAHA.123.030385. Epub 2023 Oct 13. PMID 37830344
- [Derived] Sleem A, Effron MB, Stebbins A, Wruck LM, Marquis-Gravel G, Munoz D, Re RN, Gupta K, Pepine CJ, Jain SK, Girotra S, Whittle J, Benziger CP, Farrehi PM, Knowlton KU, Polonsky TS, Roe MT, Rothman RL, Harrington RA, Jones WS, Hernandez AF. Effectiveness and Safety of Enteric-Coated vs Uncoated Aspirin in Patients With Cardiovascular Disease: A Secondary Analysis of the ADAPTABLE Randomized Clinical Trial. JAMA Cardiol. 2023 Nov 1;8(11):1061-1069. doi: 10.1001/jamacardio.2023.3364. PMID 37792369
- [Derived] Shen R, Mulder H, Wruck L, Weissler EH, Robertson HR, Sharlow AG, Kripalani S, Munoz D, Effron MB, Gupta K, Girotra S, Whittle J, Benziger CP, VanWormer JJ, Polonsky TS, Rothman RL, Harrington RA, Hernandez AF, Jones WS. Internet Versus Noninternet Participation in a Decentralized Clinical Trial: Lessons From the ADAPTABLE Study. J Am Heart Assoc. 2023 Jul 4;12(13):e027899. doi: 10.1161/JAHA.122.027899. Epub 2023 Jun 22. PMID 37345815
- [Derived] Weissler EH, Stebbins A, Wruck L, Munoz D, Gupta K, Girotra S, Whittle J, Benziger CP, Polonsky TS, Bradley SM, Hammill BG, Merritt JG, Zemon DN, Hernandez AF, Jones WS. Outcomes among patients with peripheral artery disease in the Aspirin Dosing: A Patient-Centric Trial Assessing Benefits and Long-Term Effectiveness (ADAPTABLE) study. Vasc Med. 2023 Apr;28(2):122-130. doi: 10.1177/1358863X231154951. PMID 37025023
- [Derived] O'Brien EC, Mulder H, Jones WS, Hammill BG, Sharlow A, Hernandez AF, Curtis LH. Concordance Between Patient-Reported Health Data and Electronic Health Data in the ADAPTABLE Trial. JAMA Cardiol. 2022 Dec 1;7(12):1235-1243. doi: 10.1001/jamacardio.2022.3844. PMID 36322059
- [Derived] Marquis-Gravel G, Faulkner M, Merritt G, Farrehi P, Zemon N, Robertson HR, Jones WS, Kraschnewski J. Importance of patient engagement in the conduct of pragmatic multicenter randomized controlled trials: The ADAPTABLE experience. Clin Trials. 2023 Feb;20(1):31-35. doi: 10.1177/17407745221118559. Epub 2022 Aug 23. PMID 35999816
- [Derived] Jones WS, Mulder H, Wruck LM, Pencina MJ, Kripalani S, Munoz D, Crenshaw DL, Effron MB, Re RN, Gupta K, Anderson RD, Pepine CJ, Handberg EM, Manning BR, Jain SK, Girotra S, Riley D, DeWalt DA, Whittle J, Goldberg YH, Roger VL, Hess R, Benziger CP, Farrehi P, Zhou L, Ford DE, Haynes K, VanWormer JJ, Knowlton KU, Kraschnewski JL, Polonsky TS, Fintel DJ, Ahmad FS, McClay JC, Campbell JR, Bell DS, Fonarow GC, Bradley SM, Paranjape A, Roe MT, Robertson HR, Curtis LH, Sharlow AG, Berdan LG, Hammill BG, Harris DF, Qualls LG, Marquis-Gravel G, Modrow MF, Marcus GM, Carton TW, Nauman E, Waitman LR, Kho AN, Shenkman EA, McTigue KM, Kaushal R, Masoudi FA, Antman EM, Davidson DR, Edgley K, Merritt JG, Brown LS, Zemon DN, McCormick TE 3rd, Alikhaani JD, Gregoire KC, Rothman RL, Harrington RA, Hernandez AF; ADAPTABLE Team. Comparative Effectiveness of Aspirin Dosing in Cardiovascular Disease. N Engl J Med. 2021 May 27;384(21):1981-1990. doi: 10.1056/NEJMoa2102137. Epub 2021 May 15. PMID 33999548
- [Derived] Ahmad FS, Ricket IM, Hammill BG, Eskenazi L, Robertson HR, Curtis LH, Dobi CD, Girotra S, Haynes K, Kizer JR, Kripalani S, Roe MT, Roumie CL, Waitman R, Jones WS, Weiner MG. Computable Phenotype Implementation for a National, Multicenter Pragmatic Clinical Trial: Lessons Learned From ADAPTABLE. Circ Cardiovasc Qual Outcomes. 2020 Jun;13(6):e006292. doi: 10.1161/CIRCOUTCOMES.119.006292. Epub 2020 May 29. PMID 32466729
- [Derived] Marquis-Gravel G, Roe MT, Robertson HR, Harrington RA, Pencina MJ, Berdan LG, Hammill BG, Faulkner M, Munoz D, Fonarow GC, Nallamothu BK, Fintel DJ, Ford DE, Zhou L, Daugherty SE, Nauman E, Kraschnewski J, Ahmad FS, Benziger CP, Haynes K, Merritt JG, Metkus T, Kripalani S, Gupta K, Shah RC, McClay JC, Re RN, Geary C, Lampert BC, Bradley SM, Jain SK, Seifein H, Whittle J, Roger VL, Effron MB, Alvarado G, Goldberg YH, VanWormer JL, Girotra S, Farrehi P, McTigue KM, Rothman R, Hernandez AF, Jones WS. Rationale and Design of the Aspirin Dosing-A Patient-Centric Trial Assessing Benefits and Long-term Effectiveness (ADAPTABLE) Trial. JAMA Cardiol. 2020 May 1;5(5):598-607. doi: 10.1001/jamacardio.2020.0116. PMID 32186653
- See also: ADAPTABLE public website — http://theaspirinstudy.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ASA 81mg | ASA 325mg
Started | 7540 | 7536
Completed | 6962 | 6828
Not Completed | 578 | 708
Not completed — Death | 357 | 315
Not completed — Withdrawal by Subject | 221 | 393

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASA 81mg | ASA 325mg | Total
Number analyzed (Participants) | 7540 | 7536 | 15076
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 66.9 [60.7 to 73.6] | 66.8 [60.37 to 73.5] | 66.8 [60.7 to 73.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2307 | 2417 | 4724
  Male | 5233 | 5119 | 10352
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 249 | 232 | 481
  Not Hispanic or Latino | 6816 | 6737 | 13553
  Unknown or Not Reported | 475 | 567 | 1042
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 69 | 45 | 114
  Asian | 82 | 64 | 146
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 664 | 647 | 1311
  White | 6014 | 5976 | 11990
  More than one race | 71 | 63 | 134
  Unknown or Not Reported | 640 | 741 | 1381

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing All-cause Death, Hospitalization for Nonfatal MI, or Hospitalization for Nonfatal Stroke in High-risk Patients With a History of MI or Documented Atherosclerotic Cardiovascular Disease (ASCVD)
Time Frame: Time of randomization through study completion, approximately 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | ASA 81mg | ASA 325mg
Number analyzed (Participants) | 7434 | 7330
Participants | 590 | 569

2. Secondary Outcome: Number of Participants Experiencing All-cause Death
Time Frame: Time of randomization through study completion, approximately 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | ASA 81mg | ASA 325mg
Number analyzed (Participants) | 7434 | 7330
Participants | 315 | 357

3. Secondary Outcome: Number of Participants Experiencing Hospitalization for Nonfatal MI
Time Frame: Time of randomization through study completion, approximately 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | ASA 81mg | ASA 325mg
Number analyzed (Participants) | 7434 | 7330
Participants | 228 | 213

4. Secondary Outcome: Number of Participants Experiencing Hospitalization for Nonfatal Stroke
Time Frame: Time of randomization through study completion, approximately 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | ASA 81mg | ASA 325mg
Number analyzed (Participants) | 7434 | 7330
Participants | 102 | 92

5. Secondary Outcome: Number of Participants Requiring Coronary Revascularization Procedures (Percutaneous Coronary Intervention [PCI] or Coronary Artery Bypass Grafting [CABG])
Time Frame: Time of randomization through study completion, approximately 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | ASA 81mg | ASA 325mg
Number analyzed (Participants) | 7434 | 7330
Participants | 471 | 446

6. Secondary Outcome: Quality of Life and Functional Status, as Measured on a 5-point Scale
Description: Quality of life measures are based on an ordinal scale from 1-5, where 1 corresponds to the best outcome and 5 to the worst. Model-based mean score estimates are obtained from mixed models of each quality of life measure.
Time Frame: 2 years
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ASA 81mg | ASA 325mg
Number analyzed (Participants) | 7540 | 7536
score on a scale
  Describe Current Health | 2.77 (.011) | 2.8 (.011)
  Able to Run Errands and Shop | 1.65 (.011) | 1.66 (.012)
  In the past 7 Days, Felt Depressed | 1.69 (.010) | 1.7 (.011)
  In the past 7 Days, Felt Fatigued | 2.25 (.012) | 2.27 (.012)
  In the past 7 Days, Problems with Sleep | 2.06 (.012) | 2.10 (.012)
  Trouble doing Regular Activities | 1.84 (.012) | 1.88 (.012)
  In the past 7 Days, Pain interfered | 2.06 (.013) | 2.02 (.013)

7. Other Pre Specified Outcome: Number of Participants Experiencing Hospitalization for Major Bleeding Complications With an Associated Blood Product Transfusion
Time Frame: Time of randomization through study completion, approximately 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | ASA 81mg | ASA 325mg
Number analyzed (Participants) | 7434 | 7330
Participants | 53 | 44

ADVERSE EVENTS:
Time Frame: Up to 50 months
Arm/Group | ASA 81mg | ASA 325mg
All-Cause Mortality (participants affected / at risk) | 315/7434 | 357/7330
Serious Adverse Events (participants affected / at risk) | 383/7434 | 349/7330
Other Adverse Events (participants affected / at risk) | 491/7434 | 471/7330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASA 81mg (N=7434) | ASA 325mg (N=7330)
Non-Fatal MI (Cardiac disorders) | 228 (228) | 213 (213)
Non-Fatal Stroke (Vascular disorders) | 102 (102) | 92 (92)
Major Bleeding (Cardiac disorders) | 53 (53) | 44 (44) — Major Bleeding requiring transfusion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASA 81mg (N=7434) | ASA 325mg (N=7330)
PCI or CABG (Cardiac disorders) | 471 (471) | 446 (446)
Transient ischemia attack (TIA) (Cardiac disorders) | 20 (20) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT02697916/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT02697916/SAP_001.pdf